CLINICAL TRIAL: NCT04252833
Title: Open-label, Crossover, Food Effect Study to Evaluate the Single Dose Pharmacokinetics of CT-044, a Reactive Species Decomposition Accelerant, in Healthy Human Volunteers
Brief Title: Open-label, Crossover, Food Effect Study to Evaluate CT-044 in Healthy Human Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lotus Clinical Research, LLC (Other)
Collaborators: CerSci Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT044-003
Record Dates: First submitted 2019-12-03; First posted 2020-02-05 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Pain, Acute; Acute Pain; Surgery; Neuropathy
Keywords: Safety; Tolerability; Single Dose; Pharmacokinetics; PK; CT-044 HCl; Food Effect
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: The dose to be utilized for the evaluation of food effect will be CT-044 600 mg single dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CT-044 600 mg (Experimental): The dose to be utilized for the evaluation of food effect will be CT-044 600 mg single dose.
  Interventions: Drug: CT-044

INTERVENTIONS:
Drug: CT-044 — CT-044 HCl is a reactive species decomposition accelerant

SUMMARY:
This open-label study will be conducted to assess the bioavailability and PK of oral single doses of CT-044 following administration with and without food and to evaluate the safety and tolerability of CT-044 when given with and without food.

DETAILED DESCRIPTION:
The food effect study will be an open-label, 2-sequence, balanced crossover design in 12 subjects previously untreated with CT-044.

Eligible subjects will be admitted to the Clinical Trial Unit on the day prior to dosing and remain in house until Day 3. Each subject will receive CT-044 single oral dose once under fed conditions (i.e., a high fat meal per FDA recommendations) and once in the fasted state.

9 Subjects will return to the Clinical Trial Unit on an outpatient basis for follow-up. Subjects will return to the Clinical Trial Unit to be treated by the second sequence after a washout period of at least 7 days, but no more than 14 days. All procedures will be repeated for the second treatment sequence. When possible, the procedures conducted at the 144-hour follow-up visit for the first sequence may serve as baseline for the second sequence of the crossover.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 through 55 years, inclusive.
* Body mass index within the range 18.5 to 32.0 kg/m2 (inclusive).
* Healthy subjects as determined by medical history, physical examination including neurological examination, vital signs, electrocardiogram (ECG), and clinical laboratory tests.
* Negative tests for hepatitis B surface antigen, hepatitis C virus antibodies and human immunodeficiency virus (HIV-1 or HIV-2) antibody, and syphilis at screening.
* Nonsmokers or ex-smokers and agrees not to use nicotine containing products from screening through 48 hours after final discharge from the Clinical Trial Unit.
* Negative screen for alcohol and drugs of abuse at screening and admission.
* Women must not be of childbearing potential by reason of surgery or at least 1 year postmenopausal (i.e., 12 months without menstrual period), or menopause confirmed with an estradiol level of <30 pg/mL and follicle-stimulating hormone level of >40 IU/L at screening.
* Men must be infertile, or truly abstinent of heterosexual intercourse, or heterosexual partner is not of childbearing potential, or must agree to use an effective method of contraception throughout the study and for 28 days after last dose of study drug. Men must agree to not provide sperm donation during that same period.
* Able and willing to be available for the duration of the study.
* Willing and able to give written informed consent to participate.
* Able to understand and comply with protocol instructions.
* Agree not to receive any vaccination within 21 days prior to admission and through Day 7 after final discharge from the Clinical Trial Unit.
* Agrees not to use nonprescription drugs, including vitamins, antacids, and herbal and dietary supplements within 14 days or 5 drug elimination half-lives, whichever is longer.

Exclusion Criteria:

- Subjects with significant previous or ongoing disease or disorder, including for example: cardiovascular diseases; hypertension; cancer or neoplasia; diabetes; hepatic, endocrine, metabolic, respiratory, renal, gastrointestinal (except appendectomy), hematological or Axis I or II psychiatric disorders.

* Clinical laboratory test results outside the normal range at screening that are considered clinically significant by the Investigator.
* Clinically significant, in the opinion of the Investigator, infection or inflammation at time of screening or admission.
* Acute gastrointestinal symptoms at time of screening or admission or a clinical diagnosis of irritable bowel syndrome (IBS) per ROME IV criteria.
* Average QTcF interval recorded on screening and pre-dose ECG must be not more than 450 msec.
* Any current or previous illicit use of Class A drugs such as opiates, cocaine, ecstasy, lysergic acid diethylamide (LSD), and amphetamines (Class B).
* An alcoholic intake greater than 14 units per week or unwillingness to stop alcohol consumption for the duration of the study.
* Use of any investigational medication within 3 months prior to the start of this study or scheduled to receive an investigational drug during the course of this study, or for 30 days or five half-lives, whichever is longer, following the last dose of study medication.
* History of severe allergies or multiple adverse drug reactions, including penicillin and cephalosporins.
* Any condition which compromises their ability to give informed consent or to communicate with the Investigator as required for the completion of this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Comparison of the maximum drug concentration | 7 days
  Following administration with and without food (Cmax) of oral single dose of CT-044
Comparison of the Time of maximum drug concentration (tmax) | 7 days
  Following a single oral dose of CT-044 following administration with and without food
Comparison of the Area under the drug concentration Time curve from time 0 extrapolated to infinity (AUC0-∞) | 7 days
  Following a single oral dose of CT-044 following administration with and without food
Comparison of the Area under the drug concentration Time curve from time 0 to the time of the last quantifiable concentration (AUC0-last) | 7 days
  Following a single oral dose of CT-044 following administration with and without food
Comparison of the Apparent oral clearance (CL/F) | 7 days
  Following a single oral dose of CT-044 following administration with and without food
Comparison of the Apparent volume distribution (Vz/F) | 7 days
  Following a single oral dose of CT-044 following administration with and without food
Comparison of the Terminal half-life (t1/2) | 7 days
  Following a single oral dose of CT-044 following administration with and without food
Comparison of the Terminal rate constant (λz) | 7 days
  Following a single oral dose of CT-044 following administration with and without food
Comparison of the Relative bioavailability | 7 days
  Following a single oral dose of CT-044 after administration of a high-fat meal (F)
Peak Plasma Concentration (Cmax) | 7 days
  Linear mixed model appropriate for a 2-period cross-over design with fixed terms for sequence, period and food condition will be used to investigate the food interaction on the Peak Plasma Concentration (Cmax)
Plasma concentration versus time curve (AUC) | 7 days
  Linear mixed model appropriate for a 2-period cross-over design with fixed terms for sequence, period and food condition will be used to investigate the food interaction Area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Lotus Clinical Resarch,LLC, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Squillace S, Salvemini D. Nitroxidative stress in pain and opioid-induced adverse effects: therapeutic opportunities. Pain. 2022 Feb 1;163(2):205-213. doi: 10.1097/j.pain.0000000000002347. No abstract available. PMID 34145168